CLINICAL TRIAL: NCT04350736
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, Sponsor-open, SAD and MAD Study in Healthy Subjects to Evaluate the Safety, Tolerability, and PK of Inhaled TD-0903, a Potential Treatment for ALI Associated With COVID-19
Brief Title: First in Human SAD and MAD Study of Inhaled TD-0903, a Potential Treatment for ALI Associated With COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 0183; 2020-000577-24 (EudraCT Number)
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Acute Lung Injury (ALI) Associated With COVID-19; Inflammatory Lung Conditions Associated With COVID-19
Keywords: Acute lung injury; ALI; COVID-19; Coronavirus Disease 2019; inflammatory lung conditions; Inflammatory lung disease
MeSH Terms: conditions — Acute Lung Injury; COVID-19 | interventions — nezulcitinib

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TD-0903 for SAD (Part A) (Experimental): 6 out of 8 subjects per cohort (up to 3 cohorts) will be randomized to receive TD-0903
  Interventions: Drug: TD-0903
- Placebo for SAD (Part A) (Experimental): 2 out of 8 subjects per cohort (up to 3 cohorts) will be randomized to receive placebo
  Interventions: Drug: Placebo
- TD-0903 for MAD (Part B) (Experimental): 8 out of 10 subjects per cohort (up to 3 cohorts) will be randomized to receive TD-0903
  Interventions: Drug: TD-0903
- Placebo for MAD (Part B) (Experimental): 2 out of 10 subjects per cohort (up to 3 cohorts) will be randomized to receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-0903 — Study drug to be administered by inhalation
  Arms: TD-0903 for MAD (Part B); TD-0903 for SAD (Part A)
Drug: Placebo — Placebo to be administered by inhalation
  Arms: Placebo for MAD (Part B); Placebo for SAD (Part A)

SUMMARY:
This is a phase 1 study in healthy subjects to evaluate the safety, tolerability and pharmacokinetics of single (Part A and B) and multiple (Part B) doses of inhaled TD-0903.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at Screening and weighs at least 50 kg.
* Medically healthy with no clinically significant medical history, physical examination, spirometry, vital signs or ECGs.
* Forced expiratory volume in 1 second (FEV1) ≥80%.
* No clinically significant abnormalities in the results of laboratory evaluations.
* Female subjects must be either of non-childbearing potential or if of childbearing potential, subject must not be pregnant or breastfeeding, and must agree to use a highly effective birth control method.
* Male subjects must agree to use condoms, in addition to the use of highly effective pregnancy prevention measures with female partners of childbearing potential.
* Understands the correct technique for the use the nebulizer device(s).
* Other inclusion criteria apply

Exclusion Criteria:

* History or presence of clinically significant medical or psychiatric condition.
* Abnormal ECG measurements at Screening.
* Any signs of respiratory tract infection within 6 weeks of Screening.
* Subject who has a current bacterial, parasitic, fungal, or viral infection; any infection requiring hospitalization or intravenous antibiotics within 6 months prior to Screening.
* Positive test for SARS-CoV-2
* Subject has any condition of the oro-laryngeal or respiratory tract.
* Uses or has used tobacco or nicotine-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, patches etc.) within 6 months prior to screening
* Additional exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of SAD of TD-0903: Adverse Events | Day 1 to Day 8
  Number and severity of treatment emergent adverse events
Safety and Tolerability of MAD of TD-0903: Adverse Events | Day 1 to Day 14
  Number and severity of treatment emergent adverse events

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of TD-0903 when given as a Single Ascending Dose (SAD): AUC | Day 1 through Day 4
  Multiple PK variables of TD-0903 will be assessed during SAD and may include, but are not limited to: Area under the plasma concentration-time curve (AUC)
Pharmacokinetics (PK) of TD-0903 when given as a Single Ascending Dose (SAD): Cmax | Day 1 through Day 4
  Multiple PK variables of TD-0903 will be assessed during SAD and may include, but are not limited to: Maximum observed concentration (Cmax)
Pharmacokinetics (PK) of TD-0903 when given as a Single Ascending Dose (SAD): Tmax | Day 1 through Day 4
  Multiple PK variables of TD-0903 will be assessed during SAD and may include, but are not limited to: Time to reach maximum observed concentration (Tmax)
Pharmacokinetics (PK) of TD-0903 when given as a Multiple Ascending Dose (MAD): AUC | Day 1 through Day 9
  Multiple PK variables of TD-0903 will be assessed during MAD and may include, but are not limited to: Area under the plasma concentration-time curve (AUC)
Pharmacokinetics (PK) of TD-0903 when given as a Multiple Ascending Dose (MAD): Cmax | Day 1 through Day 9
  Multiple PK variables of TD-0903 will be assessed during MAD and may include, but are not limited to: Maximum observed concentration (Cmax)
Pharmacokinetics (PK) of TD-0903 when given as a Multiple Ascending Dose (MAD): Tmax | Day 1 through Day 9
  Multiple PK variables of TD-0903 will be assessed during MAD and may include, but are not limited to: Time to reach maximum observed concentration (Tmax)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Theravance Biopharma Investigational Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.